CLINICAL TRIAL: NCT01365611
Title: Open Label Study to Assess the Pharmacokinetics of Intranasal Ketorolac Tromethamine Following Multiple Doses of Fluticasone Propionate in Healthy Subjects
Brief Title: Open Label Study to Assess the Pharmacokinetics of Intranasal Ketorolac Tromethamine Following Fluticasone Propionate in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egalet Ltd (Industry)
Responsible Party: David Bregman, M.D., Ph.D., Luitpold Pharmaceuticals, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROX 2006-04
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Results first posted 2013-04-30 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-02

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Ketorolac Tromethamine; Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ketorolac tromethamine (Experimental)
  Interventions: Drug: Ketorolac tromethamine; Drug: Fluticasone Propionate

INTERVENTIONS:
Drug: Ketorolac tromethamine — A single intranasal dose of 30 mg ketorolac tromethamine was administered to all subjects on Days 1 and 6.
Drug: Fluticasone Propionate — Daily intranasal dose of 200 ug fluticasone propionate on Days 2-6

SUMMARY:
This was a non-randomized, open label study in healthy male and female volunteers. A single intranasal dose of 30 mg ketorolac tromethamine was administered to all subjects on Days 1 and 6; in addition, subjects received a daily intranasal dose of 200 µg fluticasone propionate on Days 2-6. Subjects remained resident in the Clinical Unit from the evening of Day 1 until the morning of Day 2 and from the evening of Day 5 until the morning of Day 7, and made ambulatory visits to the Clinical Unit on the morning of Days 3-5. A post study medical was performed within 7 days of study completion.

The objective of this study was to assess the effects of chronic administration of fluticasone propionate on the pharmacokinetics of intranasal ketorolac in healthy male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers aged 18 to 60 years inclusive
* Female subjects of child bearing potential must have had a negative urine pregnancy test prior to entry into the study and must not have been breastfeeding
* All male subjects with female partners of child bearing potential must have consented to use a medically acceptable method of contraception (oral or implanted contraceptive hormones, intrauterine device or surgical sterilization plus condom or diaphragm with spermicidal agent) throughout the study period
* Subject must have given signed informed consent
* Subject was within 20% of the normal weight for his/her height and body build according to the table of "Desirable Weights for Men and Women" (Metropolitan Life Insurance Co. 1999)
* Subject's medical history was considered normal, with no clinically significant abnormalities
* Subject was considered to be in good health in the opinion of the Investigator as determined by a pre-study physical examination with no clinically significant abnormalities, vital signs within normal ranges and an electrocardiogram (ECG) with no clinically significant abnormalities
* Subject's pre study clinical laboratory findings were within the normal range or if outside of the normal range were not deemed clinically significant in the opinion of the Investigator
* Subject had bilateral patent nasal airways at screening and Day 1 as assessed by the Investigator
* Subject had a body weight of at least 60 kg

Exclusion Criteria:

* Subject had had a clinically significant illness in the 4 weeks before screening
* Subject had used prescribed medications in the 3 weeks prior to dosing or over-the-counter preparations for 7 days prior to dosing, except paracetamol which was allowed up to 48 h prior to dosing. However, use of multivitamins and oral contraceptives was permitted
* Subject had a significant history of drug/solvent abuse, or a positive drugs of abuse (DOA) test at screening
* Subject had a history of alcohol abuse or currently drank in excess of 28 units per week (males) or 21 units per week (females)
* Subject was a current user of tobacco or had a history of smoking in the past 5 years
* Subject was in the opinion of the Investigator not suitable to participate in the study
* Subject had participated in any clinical study with an investigational drug/device within 3 months prior to dosing
* Subject had a positive result of human immunodeficiency virus (HIV) screen, hepatitis B screen or hepatitis C screen
* Subject had had a serious adverse reaction or significant hypersensitivity to any drug
* Subject had donated 500 mL or more of blood within the 3 months prior to screening
* Subject had any history of co-existing nasal polyps, nonsteroidal anti-inflammatory drug (NSAID) sensitivity and asthma
* Subject had had an allergic reaction to aspirin or other NSAIDs
* Subject had a current upper respiratory tract infection or other respiratory tract condition that could interfere with the absorption of the nasal spray or with the assessment of adverse events (AEs)
* Any suspicion of rhinitis medicamentosa (chronic daily use of topical decongestants)
* Subject had used a monoamine oxidase inhibitor in the 14 days prior to study entry
* Subject had active peptic ulcer disease, gastrointestinal bleeding or perforation, or a history of peptic ulcer disease or gastrointestinal bleeding
* Subject had anemia due to unexplained or known gastrointestinal bleeding
* Subject had a history of asthma or any other chronic pulmonary disorder
* Subject had renal impairment or a risk of renal failure due to volume depletion
* Subject had a previous history of nasal surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-02; Primary Completion 2007-05 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cyril Clarke, BSc MB BS MFPM, Principal Investigator — ICON Development Solutions
Locations (1):
- ICON Development Solutions, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: February 7, 2007 - May 22, 2007; Clinical Unit
Groups:
- All Study Participants: A single intranasal dose of 30 mg ketorolac tromethamine was administered to all subjects on Days 1 and 6.
  Subjects received a single daily intranasal dose of 200mg fluticasone propionate on Days 2-6 followed by a single intranasal dose of 30mg ketorolac tromethamine administered 30 minutes after fluticasone propionate on Day 6.
Period: Overall Study
Arm/Group | All Study Participants
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 35
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 26
Region of Enrollment [Number; unit: participants]
  United Kingdom | 36

OUTCOME MEASURES:

1. Primary Outcome: Cmax (the Maximum Observed Plasma Concentration of Ketorolac Tromethamine)
Time Frame: PK parameters were determined using the following blood sampling times: pre-dose (within 10 minutes of ketorolac tromethamine administration), 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 15 and 24 h post administration of study drug on Days 1 and 6
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Ketorolac Tromethamine (Given Alone): A single intranasal dose of 30 mg ketorolac tromethamine was administered to all subjects on Days 1 and 6.
- Fluticasone Propionate + Ketorolac Tromethamine: Subjects received a single daily intranasal dose of 200mg fluticasone propionate on days 2-6 followed by a single intranasal dose of 30mg ketorolac tromethamine administered 30 minutes after fluticasone propionate on Day 6.
Arm/Group | Ketorolac Tromethamine (Given Alone) | Fluticasone Propionate + Ketorolac Tromethamine
Number analyzed (Participants) | 36 | 36
ng/mL | 2128 (1042.5) | 1948 (1018.3)

2. Primary Outcome: Tmax (the Time to Maximum Concentration of Ketorolac Tromethamine)
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Ketorolac Tromethamine (Given Alone) | Fluticasone Propionate + Ketorolac Tromethamine
Number analyzed (Participants) | 36 | 36
hours | 0.750 [0.25 to 1.00] | 0.750 [0.25 to 1.00]

3. Primary Outcome: AUC 0-t (the Area Under the Plasma Concentration-time Curve (AUC) From Time Zero to the Last Quantifiable Time Point Post-dose of Ketorolac Tromethamine).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hours/mL
Arm/Group | Ketorolac Tromethamine (Given Alone) | Fluticasone Propionate + Ketorolac Tromethamine
Number analyzed (Participants) | 36 | 36
ng*hours/mL | 7991 (4364.2) | 7610 (4076.8)

4. Primary Outcome: AUC Inf (the AUC From Time Zero to Infinity, Where Possible)
Time Frame: as for outcome 1
Population: The half-life could not be estimated for a subject due to the nature of the subject's PK profile.
Measure: Mean (Standard Deviation); unit: ng*hours/mL
Arm/Group | Ketorolac Tromethamine (Given Alone) | Fluticasone Propionate + Ketorolac Tromethamine
Number analyzed (Participants) | 35 | 36
ng*hours/mL | 8970 (4575) | 8276 (4380.7)

5. Primary Outcome: t1/2z (the Terminal Half-life of Ketorolac Tromethamine, Where Possible)
Time Frame: as for outcome 1
Population: The half-life could not be estimated for a subject due to the nature of the subject's PK profile.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ketorolac Tromethamine (Given Alone) | Fluticasone Propionate + Ketorolac Tromethamine
Number analyzed (Participants) | 35 | 36
hours | 5.95 (2.105) | 5.49 (2.004)

6. Primary Outcome: MRT (the Mean Residence Time of Ketorolac Tromethamine, Where Possible)
Time Frame: as for outcome 1
Population: The half-life could not be estimated for a subject due to the nature of the subject's PK profile.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ketorolac Tromethamine (Given Alone) | Fluticasone Propionate + Ketorolac Tromethamine
Number analyzed (Participants) | 35 | 36
hours | 7.05 (2.141) | 6.53 (2.354)

ADVERSE EVENTS:
Time Frame: 3 months and 2 weeks
Arm/Group | Ketorolac Tromethamine (Given Alone) | Fluticasone Propionate + Ketorolac Tromethamine
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 8/36 | 7/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketorolac Tromethamine (Given Alone) (N=36) | Fluticasone Propionate + Ketorolac Tromethamine (N=36)
Fatigue (General disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 4 (5) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 4 (4)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No